CLINICAL TRIAL: NCT05780255
Title: Quality of Life 1y and 2 y After VV-ECMO for COVID-19, Measured by the 36-item Short Form Health Survey
Brief Title: Quality of Life 1y and 2 y After VV-ECMO for COVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-19-ECMO BC-09806
Record Dates: First submitted 2023-03-13; First posted 2023-03-22 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; Extracorporeal Membrane Oxygenation Complication; Quality of Life; Death
Keywords: ECMO; COVID-19; quality of life
MeSH Terms: conditions — Death; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 positive patients: Patients with a PCR-confirmed COVID-19 infection, with ARDS and supported by VV-ECMO
  Interventions: Device: VV-ECMO

INTERVENTIONS:
Device: VV-ECMO — veno-venous extracorporeal membrane oxygenation

SUMMARY:
This study aims to investigate the quality of life and the outcome after veno-venous extracoporeal membrane oxygenation (ECMO) support fir severe acute respiratory syndrome (ARDS) in COVID-19 patients.

DETAILED DESCRIPTION:
The investigators follow our COVID-19 patients supported by ECMO, we make phone calls or real-life visits to pthe patients to score the quality of life, by using the SF-36. The SF-36 measures eight scales: physical functioning, role physical, bodily pain, general health, vitality , social functioning , role emotional , and mental health.

The participants are contacted 3 months, 6months, 1year and 2 years after the ECMO support started for evaluation of the SF-36.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PCR-confirmed COVID-19 infection AND
* Acute Respiratory Distress Syndrome who require veno-venous ECMO therapy.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PCR-confirmed COVID-19 infection with ARDS who require veno-venous ECMO therapy.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
in-hospital mortality | mortality during hospitalisation, up to two years
Quality of life 1y after ECMO insertion | 1 year
  Result of SF-36 1 year after VV-ECMO insertion
Quality of life 2y after ECMO insertion | 2 years
  Result of SF-36 2 years after VV-ECMO insertion

SECONDARY OUTCOMES:
Lung complications requiring surgical treatment | From the start of VV-ECMO support until weaning of VV-ECMO, up to two years
  Hemothorax or lung abcedation
Duration of mechanical ventilation | 2 years
LOS ICU | from the day of intensive care unit admission until the day of transfer to the ward, up to two years
  length of stay at the intensive care unit
LOS hospital | from the day of hospital admission until the day that the participant is transferred to home, up to two years
  length of stay at the hospital
death after hospital discharge | after discharge from the hospital upon 2 years after
  all-cause death
Incidence of acute kidney injury | from the day of hospital admission until the day that the participant is transferred to home, up to two years

CONTACTS AND LOCATIONS:
Overall Officials: Harlinde Peperstraete, Principal Investigator — UZ Gent
Locations (1):
- Ghent university hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No